CLINICAL TRIAL: NCT02432183
Title: Longitudinal Follow-up of Exercise-induced Bronchoconstriction and Airway Inflammation in High School Athletes
Brief Title: Longitudinal Follow-up of High School Athletes
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dominque Bullens, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S53448
Record Dates: First submitted 2015-03-27; First posted 2015-05-04 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Elite Athlete; Healthy
Keywords: individual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — induced sputum sample and venous blood (serum)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Football players: Football players of the first grade of high school are recruited from the topsportschool in Leuven.
- Basketball players: Basketball players of the first grade of high school are recruited from the topsportschool in Leuven.
- Swimmers: Swimmers of the first grade of high school are recruited from the future team of the Flemish Swimming Federation
- Control group: Age-matched controls are recruited (exercising at a recreational level, >4 hours).

SUMMARY:
In this study the investigators will study the lung function and airway inflammation in elite athletes starting at the elite sport school (age: 12-13 year) and the change in lung function parameters and airway inflammation after 1 and 2 years at the elite sport school in comparison to age-matched controls (exercising at a recreational level, <4 hours/week).

DETAILED DESCRIPTION:
A group of elite athletes (from the elite sport school in Leuven (n=35) in cooperation with 'Sportmedisch Advies Centrum' (SMAC) UZ Leuven) and the future team of the Flemish Swimming Federation (n=15) will be recruited at the start of their career (first level) as an elite athlete. A group of healthy subjects (n=20) will be recruited to serve as a control.

The investigators will compare lung function parameters and airway inflammation at the first visit in the autumn of 2011 and the second and third visit (one and two years later, respectively).

Lung function will be assessed by spirometry. Sputum will be induced with an aerosol of inhaled hypertonic saline in concentrations of 3%, 4% and 5% for 7 minutes generated by a De Vilbiss nebuliser (Ultra-Neb 2000 model 200HI) after pretreatment with 400 mg inhaled salbutamol. Sputum will be processed as previously described and the obtained cell suspensions will be used for differential cell counts and cytokine mRNA analysis. The supernatant will be used to measure cytokine and chemokine levels.

EIA diagnosis (visit 1,2 and 3) will be assessed by a diagnostic test for asthma (positive reversibility test with salbutamol) and a positive EIB-test. Eucapnic voluntary hyperventilation test will be used as a test for EIB (gold standard of IOC-MC). Dynamic lung function parameters will be assessed before and immediately after, 5' after, 10' after and 15' after eucapnic hyperventilation. Patients were asked to breath at 85% of the maximal ventilation (predefined as maximal voluntary volume) for 6 minutes through a mouthpiece connected to a reservoir. The reservoir is be filled with a gas mixture of 21% 02, 5% CO2 and 74% N2. The test is considered positive when a drop in FEV1 of >10% occurred at one of the time points after eucapnic hyperventilation.

ELIGIBILITY:
Inclusion Criteria:

* Elite athletes from the elite sport school in Wilrijk and Leuven
* First grade of high school

Exclusion Criteria:

* Performing >4hours/week sports

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A group of elite athletes at the start of their career (both from the elite sport school in Wilrijk (n=15) and Leuven (n=35) in cooperation with 'Sportmedisch Advies Centrum' (SMAC) UZ Leuven) are recruited. Three sport disciplines are included: basketball players, football players and swimmers.
  A group of healthy subjects (n=20) is recruited to serve as a control.
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

REFERENCES:
- [Background] Bonini M, Braido F, Baiardini I, Del Giacco S, Gramiccioni C, Manara M, Tagliapietra G, Scardigno A, Sargentini V, Brozzi M, Rasi G, Bonini S. AQUA: Allergy Questionnaire for Athletes. Development and validation. Med Sci Sports Exerc. 2009 May;41(5):1034-41. doi: 10.1249/MSS.0b013e318193c663. PMID 19346984
- [Result] Van der Eycken S, Schelpe A, Marijsse G, Dilissen E, Troosters T, Vanbelle V, Aertgeerts S, Dupont LJ, Peers K, Bullens DM, Seys SF. Feasibility to apply eucapnic voluntary hyperventilation in young elite athletes. Respir Med. 2016 Feb;111:91-3. doi: 10.1016/j.rmed.2015.12.012. Epub 2016 Jan 4. PMID 26790574
- [Result] Jonckheere AC, Seys SF, Dilissen E, Marijsse G, Schelpe AS, Van der Eycken S, Verhalle T, Vanbelle V, Aertgeerts S, Troosters T, Peers K, Dupont LJ, Bullens DMA. AQUA(c) Questionnaire as prediction tool for atopy in young elite athletes. Pediatr Allergy Immunol. 2018 Sep;29(6):648-650. doi: 10.1111/pai.12949. Epub 2018 Jul 9. No abstract available. PMID 29908073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: total number of control subjects is increased compared to protocol enrollment to compensate for gender imbalance
Pre-assignment Details: As we did not anticipate a gender imbalance in the study groups, control subjects were recruited based on age-match not on sex-match. To correct for the gender imbalance, we added nine control subjects to the control group.
Period: Overall Study
Arm/Group | Football Players | Swimmers | Basketball Players | Control Group
Started | 44 | 47 | 26 | 17
Completed | 44 | 47 | 26 | 17
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Football Players | Swimmers | Basketball Players | Control Group | Total
Number analyzed (Participants) | 44 | 47 | 26 | 17 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44 | 47 | 26 | 17 | 134
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.1 (0.9) | 12.1 (0.8) | 12.2 (0.6) | 12.9 (1.8) | 12.5 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 12 | 12 | 42
  Male | 37 | 36 | 14 | 5 | 92
Region of Enrollment [Number; unit: participants]
  Belgium | 44 | 47 | 26 | 17 | 134

OUTCOME MEASURES:

1. Primary Outcome: Maximal Fall in Forced Expiratory Volume in One-second (FEV1) After Eucapnic Voluntary Hyperventilation (EVH) Test
Description: percentage change in FEV1 after EHV test compared to baseline EVH test will be performed for 6 min at a target ventilation of 85% of the maximal voluntary ventilation (MVV), which will be determined before initiation of the test. Ventilation will be monitored during the 6-min test by a flow sensor (Jaeger Oxycon Mobile, Carefusion), FEV1 will be measured immediately after challenge and at 5, 10 and 15 min. A reduction in FEV1 ≥ 10% at one of the time points compared with the value before the test will be considered positive. Salbutamol (400 μg) will be given after the last spirometry (post-EVH) to check bronchodilator reversibility.
Time Frame: change from baseline compared to 15 minutes after EVH test
Population: EVH test not correctly performed (according to measure description) in 11 subjects (5 football players, 4 basket ball players and 2 swimmers) and hence 11 subjects here excluded from analysis
Measure: Median (Inter-Quartile Range); unit: percentage of change in FEV1 after EVH
Arm/Group | Football Players | Basketball Players | Swimmers | Control Group
Number analyzed (Participants) | 39 | 22 | 45 | 17
percentage of change in FEV1 after EVH | -4 [-11 to 3] | -9 [-18 to 0] | -9 [-15 to -2] | -5 [-11 to 1]
Statistical Analysis 1: Comparison: Football Players vs Basketball Players vs Swimmers vs Control Group; Test type: Superiority or Other; p = 0.0061, Kruskal-Wallis; post-hoc comparison with Dunn's multiple comparison test: p=0.0326 between arm 1 and 2; p=0.0147 between arm 1 and 3

2. Secondary Outcome: Number of Participants With Allergies Determined by Positive Skin Prick Test
Time Frame: baseline
Measure: Number; unit: participants
Arm/Group | Football Players | Basketball Players | Swimmers | Control Group
Number analyzed (Participants) | 44 | 26 | 47 | 17
participants | 14 | 6 | 19 | 4

3. Other Pre Specified Outcome: Number of Sputum Uric Acid-high Subjects (Determined by ELISA on Sputum Supernatants)
Description: number of subjets with sputum uric acid level above p90 in controls
Time Frame: baseline
Population: Sputum not available in 21 subjects due to technical issues (10 football players, 7 basket ball players, and 4 swimmers) and hence excluded from this analysis
Measure: Number; unit: participants
Arm/Group | Football Players | Basketball Players | Swimmers | Control Group
Number analyzed (Participants) | 34 | 19 | 43 | 17
participants | 15 | 15 | 26 | 3

ADVERSE EVENTS:
Arm/Group | Football Players | Swimmers | Basketball Players | Control Group
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/47 | 0/26 | 0/17
Other Adverse Events (participants affected / at risk) | 0/44 | 0/47 | 0/26 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes